CLINICAL TRIAL: NCT01132612
Title: A Multicenter Extension Trial of Subcutaneously Administered AIN457 in Participants With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: AIN457 Regimen Finding Extension Study in Participants With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2211E1; 2009-017234-51 (EudraCT Number)
Record Dates: First submitted 2010-05-19; First posted 2010-05-28 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Plaque-type Psoriasis
Keywords: Chronic plaque-type psoriasis; AIN457; dermatology; Moderate to severe chronic plaque-type psoriasis
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed-time interval regimen (Experimental): Secukinumab 150 mg subcutaneous (sc) administered at Week 1 (baseline) of the extension study and every 12 weeks thereafter
  Interventions: Drug: AIN457; Drug: Placebo
- Treatment at start of relapse regimen (Experimental): Placebo administered at Week 1 (baseline) of the extension study and every 12 weeks thereafter. If relapse, then switch to secukinumab 150 mg sc administered every 4 weeks
  Interventions: Drug: AIN457; Drug: Placebo
- Open-label (Experimental): Secukinumab 150 mg sc administered every 4 weeks
  Interventions: Drug: AIN457

INTERVENTIONS:
Drug: AIN457 — AIN457A 150 mg powder for solution
Drug: Placebo — Placebo to AIN457A 150 mg powder for solution
  Arms: Fixed-time interval regimen; Treatment at start of relapse regimen

SUMMARY:
The purpose of this study was to provide long term clinical data for the compound for the treatment of the indication of moderate to severe chronic plaque-type psoriasis.

DETAILED DESCRIPTION:
In the Proof-of-Concept study (CAIN457A2102/ NCT00669916), AIN457 was proven to be efficacious in the treatment of moderate to severe chronic plaque-type psoriasis. As a result, a phase IIb regimen finding study had been started (CAIN457A2211/NCT00941031).

The data gathered in this extension study of the core study (CAIN457A2211)was used to expand the safety database of the compound for the treatment of moderate to severe chronic plaque-type psoriasis. The participants in the extension study continued to stay on the exact same treatment regimen they were taking when completing the core study. The extension trial was first designed to provide long-term safety data of up to 100 weeks of treatment (32 weeks in the core study plus 68 weeks in the extension study (part 1)), and an additional 12 weeks of treatment-free follow-up for participants who did not continue in the extension study. Amendment 2 provided an additional 156 weeks of treatment (32 weeks in the core study plus 224 weeks in the extension study, equaling 256 weeks of total treatment (part 2)), before participants entered the 12 weeks of treatment-free follow-up. Protocol Amendment 3 extended the prolongation part of the study by up to 104 additional weeks of treatment (part 3) or until the drug was commercially available in the market of the country of participation, whichever occurred first.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients who completed the core study CAIN457A2211. A patient is defined as having completed the core study if he/she completed the study up to and including visit 13 (F4) of the core study
* Patients must be able to understand and communicate with the investigator and comply with the requirement of the study and must given written, signed and dated informed consent before any study assessment is performed.
* Patients must be expected to benefit from the ongoing treatment with AIN457, as assessed by the patient and investigator
* Male patients must consent to practice reliable contraception during the study and for 16 weeks after the last dose of study drug administration Note: Due to new data available from the toxicology studies, the need for male contraception was removed.

Key Exclusion Criteria:

* Patients who experience a second consecutive full relapse at visit 13 ( week F4) of the core study CAIN457A2211
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until termination of gestation, confirmed by a positive hCG laboratory test (> 5mlU/mL)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unwilling to use effective contraception during the study and for 16 weeks after stopping treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2010-05-11 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2016-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (56):
- United States (24):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Newnan, Georgia
  - Novartis Investigative Site, Snellville, Georgia
  - Novartis Investigative Site, Champaign, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Clinton Township, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Lake Oswego, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Charlottesville, Virginia
- France (2):
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Toulouse
- Germany (13):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Kopavogur, Iceland
- Israel (3):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Japan (10):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Chitose, Hokkaido
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
- Norway (3):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants continued their regimens as assigned in CAIN457A2211 (NCT00941031) and were enrolled into one of the following: fixed time interval regimen (FI), treatment at start of relapse regimen (SR) or open-label (OL). There were no more placebo treated patients at the end of the core. Therefore, there is no placebo arm in the extension.
Period: Overall Study
Arm/Group | Fixed-time Interval Regimen | Treatment at Start of Relapse Regimen | Open-label
Started | 46 | 42 | 187
Completed | 6 | 7 | 17
Not Completed | 40 | 35 | 170
Not completed — Death | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 3
Not completed — Lost to Follow-up | 2 | 2 | 7
Not completed — Adverse Event | 5 | 2 | 15
Not completed — Withdrawal by Subject | 5 | 8 | 19
Not completed — Administrative problems | 5 | 1 | 52
Not completed — Lack of Efficacy | 23 | 22 | 73

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed-time Interval Regimen | Treatment at Start of Relapse Regimen | Open-label | Total
Number analyzed (Participants) | 46 | 42 | 187 | 275
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (13.71) | 39.9 (12.12) | 45.0 (11.78) | 43.9 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 39 | 66
  Male | 31 | 30 | 148 | 209

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Deaths
Description: Safety was assessed by frequency of adverse events including serious adverse events.
Time Frame: up to week 351
Population: Extension safety set: the extension safety set consisted of all participants who received at least one dose of study drug during the extension and had at least one post-baseline safety assessment during the extension.
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed-time Interval Regimen | Treatment at Start of Relapse Regimen | Open-label
Number analyzed (Participants) | 46 | 42 | 187
Participants
  Adverse events | 44 | 41 | 180
  Serious adverse events | 9 | 4 | 43
  Deaths | 0 | 0 | 1

2. Secondary Outcome: Number of Participants With at Least 50%, 75% or 90% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) and IGA Mod 2009 0 or 1 Response
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). The IGA scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe and 5 = very severe.
Time Frame: Extension weeks: 1, 25, 73 and 301 (too few data points were available to perform analysis at week 301)
Population: Full analysis set (FAS): The FAS, which included all participants who entered the extension and to whom study drug was assigned, was considered for the analysis. Only those participants, who had evaluable data at a given time point, were analyzed at that time point.
Measure: Number; unit: Number of participants
Arm/Group | Fixed-time Interval Regimen | Treatment at Start of Relapse Regimen | Open-label
Number analyzed (Participants) | 46 | 42 | 187
Number of participants
  Extension week 1, PASI 50: number analyzed (Participants) | 46 | 40 | 174
  Extension week 1, PASI 50 | 43 | 34 | 163
  Extension week 1, PASI 75: number analyzed (Participants) | 46 | 40 | 174
  Extension week 1, PASI 75 | 31 | 16 | 102
  Extension week 1, PASI 90: number analyzed (Participants) | 46 | 40 | 174
  Extension week 1, PASI 90 | 17 | 3 | 61
  Ext. week 1, IGA mod 2009 0 or 1: number analyzed (Participants) | 44 | 38 | 168
  Ext. week 1, IGA mod 2009 0 or 1 | 24 | 7 | 70
  Extension week 25, PASI 50: number analyzed (Participants) | 35 | 33 | 159
  Extension week 25, PASI 50 | 29 | 27 | 142
  Extension week 25, PASI 75: number analyzed (Participants) | 35 | 33 | 159
  Extension week 25, PASI 75 | 19 | 10 | 91
  Extension week 25, PASI 90: number analyzed (Participants) | 35 | 33 | 159
  Extension week 25, PASI 90 | 12 | 2 | 42
  Ext. week 25, IGA mod 2009 0 or 1: number analyzed (Participants) | 35 | 33 | 159
  Ext. week 25, IGA mod 2009 0 or 1 | 15 | 4 | 48
  Extension week 73, PASI 50: number analyzed (Participants) | 19 | 19 | 114
  Extension week 73, PASI 50 | 18 | 17 | 100
  Extension week 73, PASI 75: number analyzed (Participants) | 19 | 19 | 114
  Extension week 73, PASI 75 | 14 | 8 | 66
  Extension week 73, PASI 90: number analyzed (Participants) | 19 | 19 | 114
  Extension week 73, PASI 90 | 8 | 1 | 31
  Ext. week 73, IGA mod 2009: number analyzed (Participants) | 19 | 19 | 114
  Ext. week 73, IGA mod 2009 | 9 | 4 | 35
  Extension week 301, PASI 50: number analyzed (Participants) | 0 | 0 | 3
  Extension week 301, PASI 50 |  |  | 3
  Extension week 301, PASI 75: number analyzed (Participants) | 0 | 0 | 3
  Extension week 301, PASI 75 |  |  | 2
  Extension week 301, PASI 90: number analyzed (Participants) | 0 | 0 | 3
  Extension week 301, PASI 90 |  |  | 1
  Extension week 301, IGA mod 2009: number analyzed (Participants) | 0 | 0 | 3
  Extension week 301, IGA mod 2009 |  |  | 1

3. Secondary Outcome: Long-term Immunogenicity Assessed by the Number of Participants Developing Anti Secukinumab Antibodies During the Trial
Description: Describes the number of participants tested positive for anti-secukinumab antibodies. It refers to the number of participants who had no positive values at baseline but developed them only after start of secukinumab treatment.
Time Frame: up to week 351
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed-time Interval Regimen | Treatment at Start of Relapse Regimen | Open-label
Number analyzed (Participants) | 46 | 41 | 184
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Arm/Group | Fixed-time Interval Regimen | Treatment at Start of Relapse Regimen | Open-label
Serious Adverse Events (participants affected / at risk) | 9/46 | 4/42 | 43/187
Other Adverse Events (participants affected / at risk) | 42/46 | 35/42 | 164/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed-time Interval Regimen (N=46) | Treatment at Start of Relapse Regimen (N=42) | Open-label (N=187)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Abscess bacterial (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 4
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1
Infected dermal cyst (Infections and infestations) | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 1
Streptococcus test positive (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Bladder stenosis (Renal and urinary disorders) | 0 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed-time Interval Regimen (N=46) | Treatment at Start of Relapse Regimen (N=42) | Open-label (N=187)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 11
Dental caries (Gastrointestinal disorders) | 3 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 20
Nausea (Gastrointestinal disorders) | 3 | 3 | 12
Toothache (Gastrointestinal disorders) | 4 | 1 | 14
Vomiting (Gastrointestinal disorders) | 1 | 3 | 13
Fatigue (General disorders) | 2 | 3 | 12
Influenza like illness (General disorders) | 1 | 2 | 12
Pyrexia (General disorders) | 1 | 4 | 9
Bronchitis (Infections and infestations) | 2 | 1 | 21
Conjunctivitis (Infections and infestations) | 4 | 0 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 4 | 9
Influenza (Infections and infestations) | 4 | 2 | 14
Nasopharyngitis (Infections and infestations) | 20 | 16 | 91
Oral herpes (Infections and infestations) | 1 | 1 | 10
Pharyngitis streptococcal (Infections and infestations) | 3 | 2 | 4
Sinusitis (Infections and infestations) | 9 | 3 | 17
Tonsillitis (Infections and infestations) | 1 | 0 | 14
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 28
Urinary tract infection (Infections and infestations) | 3 | 4 | 6
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 10
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2 | 10
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0 | 6
Alanine aminotransferase increased (Investigations) | 1 | 0 | 12
C-reactive protein increased (Investigations) | 3 | 0 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 3 | 14
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 43
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 30
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 11
Dizziness (Nervous system disorders) | 3 | 0 | 4
Headache (Nervous system disorders) | 11 | 6 | 29
Anxiety (Psychiatric disorders) | 0 | 0 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 14
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 13 | 16 | 59
Hypertension (Vascular disorders) | 4 | 6 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.